CLINICAL TRIAL: NCT04026204
Title: Prospective, Observational, Single Center Trial of Reobtaining Coronary Ostia Cannulation Beyond Transcatheter Aortic Valve Stent (RE-ACCESS)
Brief Title: Reobtain Coronary Ostia Cannulation Beyond Transcatheter Aortic Valve Stent (RE-ACCESS)
Acronym: RE-ACCESS
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Marco Barbanti, Principal Investigator, University of Catania
Other Study IDs: UCatania001
Record Dates: First submitted 2019-06-12; First posted 2019-07-19 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Aortic Stenosis; Coronary Artery Disease
Keywords: TAVR; Coronary cannulation; Transcatheter aortic prosthesis
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary cannulation after TAVR: Coronary ostia cannulation after TAVR

SUMMARY:
With the upcoming expansion of transcatheter aortic valve replacement (TAVR) indications to younger patients, the feasibility of coronary ostia cannulation beyond different bioprosthesis stent is currently a matter of debate. Purpose of this study is: 1) to assess the feasibility to re-engage coronary ostia after TAVR; 2) to discover potential native anatomical or prosthesis-related features that may preclude proper coronary cannulation after TAVR.

DETAILED DESCRIPTION:
Single-center, prospective, pilot study. Aim of this study is to assess the feasibility of coronary ostia re-engagement beyond transcatheter aortic valve (TAV) stent through a transfemoral access in 300 consecutive patients undergoing transfemoral TAVR with pre-procedural computed tomography assessment available.

The possibility to selectively cannulate each coronary, the amount of time and contrast will be evaluated in each patient before and after implantation of either balloon-(SAPIEN 3) or self-expanding (Evolut R/PRO, Acurate Neo or Portico) TAVs, thus generating an internal comparator.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with severe aortic stenosis undergoing TAVR with all commercially available devices
* Availability of preprocedural aortic root evaluation by computed tomography angiography scans

Exclusion Criteria:

* TAVR in degenerated bioprostheses
* Known ostial chronic total occlusion
* Transcatheter valve not deployed in its anatomical position
* Patients with hemodynamic instability during the procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic, severe aortic stenosis who underwent TAVR
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Number of patients in whom it was possible to selectively cannulate coronary ostia after TAVR | 5 minutes
  Angiographic assessment of coronary ostia selective cannulation after TAVR

SECONDARY OUTCOMES:
Hazard ratios of factors associated with the inability to selectively cannulate coronary ostia after TAVR | 5 minutes
  Aortic root CTA measurements and prosthesis implantation-related factors associated with inability to selectively cannulate coronary ostia after TAVR at multivariate regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: Marco Barbanti, MD, Principal Investigator — University of Catania
Locations (1):
- Department of Cardiology, CAST, AU Policlinico-Vittorio Emanuele, Catania, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barbanti M, Costa G, Picci A, Criscione E, Reddavid C, Valvo R, Todaro D, Deste W, Condorelli A, Scalia M, Licciardello A, Politi G, De Luca G, Strazzieri O, Motta S, Garretto V, Veroux P, Giaquinta A, Giuffrida A, Sgroi C, Leon MB, Webb JG, Tamburino C. Coronary Cannulation After Transcatheter Aortic Valve Replacement: The RE-ACCESS Study. JACC Cardiovasc Interv. 2020 Nov 9;13(21):2542-2555. doi: 10.1016/j.jcin.2020.07.006. Epub 2020 Oct 14. PMID 33069648